CLINICAL TRIAL: NCT02801682
Title: NOBICS - NOvel BIomarker In Invasive CandidiasiS/Candida Sepsis
Acronym: NOBICS
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Robert Krause, MD, Univ.Prof.Dr., Medical University of Graz
Other Study IDs: KLI 561-B31
Record Dates: First submitted 2016-06-09; First posted 2016-06-16 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Invasive Candidiasis
MeSH Terms: conditions — Candidiasis, Invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Healthy Controls
- Invasive Candidiasis
- Bacterial Sepsis (Bacteremia)
- ICU patients without infectious disease

SUMMARY:
Invasive Candida infections are serious complications in immunocompromised patients including those undergoing treatment for cancer but occur also in patients treated in ICUs. Survival rate of invasive candidiasis is associated with early initiation of antifungal therapy (15% mortality rate for candidemic patients with antifungal therapy on day 0 related to the culture date of the first blood sample positive for yeasts compared to 41% for patients who received antifungal therapy on day 3). Up to date, no laboratory method or clinical decision rule is available for correct anticipation of invasive candidiasis which would avoid delays in appropriate antifungal therapy initiation. In clinical practice culture based methods (e.g. blood cultures) miss up to 50% of invasive candidiasis cases. Preemptive antifungal therapy is therefore often initiated in critically ill patients after Candida has been isolated from various non-sterile patient samples even without any sufficient evidence for invasive candidiasis. The disadvantages of this approach include over- and undertreatment of patients (up to 50% of candidemia cases are missed, and on the other hand 89% patients are treated unnecessarily), increased selective pressure for the development of antifungal resistance, potential risk of adverse drug reactions, and increased costs (expenses for antifungal therapy account for half of the antimicrobial medication budget in tertiary care hospitals). In addition, no survival benefit could be demonstrated by this strategy in ICU patients.

The aim of this study is to identify biological markers to anticipate or support the diagnosis of invasive candidiasis in ICU patients, to overcome current deficiencies in detection of invasive candidiasis and consequently to differentiate between Candida spp. colonization and invasive Candida infection. The investigators intend to examine time dependent courses of potential host and pathogen derived biomarkers as well as innate or acquired predispositions for invasive candidiasis; e.g. automated (1→3) ß- D- Glucan tests, DNA in serum blood samples, pathogen recognition receptors and serum markers like interleukin (IL)-1, IL-2, IL-6, IL-10, IL-12, IL-17A, IL-17F, IL-22, IL-23, Tryptophan, Kynurenine, composition of indigenous microbiota of gastrointestinal and lower respiratory tract and skin, and risk factors for invasive candidiasis like underlying diseases and treatments. The study should contribute to improved assessment of ICU patients at risk for invasive candidiasis and to improved diagnosis of invasive candidiasis in ICU patients. In clinical practice the reliable differentiation between infection and colonization will allow more targeted antifungal therapy leading to enhanced antifungal treatment initiation on the one hand (in cases of true invasive candidiasis) and to reduction of unnecessary antifungal treatments and treatment costs on the other hand.

ELIGIBILITY:
ad 1:

Inclusion Criteria:

-subjects without any evidence of current or chronic infectious diseases

Exclusion Criteria:

* Clinical or radiological or laboratory evidence of current infectious disease (temperature >38°C, elevated CRP >5mg/dl, leukocytosis >11400, elevated neutrophiles)
* antifungal therapy within 8 weeks prior to inclusion
* immunosuppressive therapy (e.g. glucocorticoids, methotrexate, azathioprin, etc)
* active haematooncological diseases
* HIV positivity

ad 2:

Inclusion criteria:

-Patients with invasive Candidias/Candida sepsis as defined in recent EORTC/MSG definitions.

Exclusion criteria:

* glucocorticoid treatment with prednisone equivalent of ≥20mg/d
* inherited neutrophil deficiency
* absolute neutrophil count of ≤500cells/mm3
* antifungal therapy within 8 weeks prior to inclusion
* immunosuppressive therapy (glucocorticoids with prednisone equivalent of ≥20mg/d, methotrexate, azathioprin etc)
* active hematooncological disease
* HIV positivity

ad 3:

Inclusion criteria:

-ICU patients with sepsis and proven bacteremia (Staph. aureus or E. coli)

Exclusion criteria:

* Antifungal therapy within 8 weeks prior to inclusion
* immunosuppressive therapy (glucocorticoids with prednisone equivalent of ≥20mg/d, methotrexate, azathioprin etc)
* active hematooncological disease HIV positivity

ad 4:

Inclusion criteria:

-ICU patients without invasive candidiasis as defined above, without bacteremia and without clinical and laboratory markers of infection(e.g. intubated and mechanically ventilated patients with stroke or CPR)

Exclusion criteria:

* Clinical or radiological or laboratory evidence of current infectious disease (temperature >38°C, elevated CRP >5mg/dl, leukocytosis >11400, elevated neutrophiles)
* antifungal therapy within 8 weeks prior to inclusion
* immunosuppressive therapy (e.g. glucocorticoids, methotrexate, azathioprin, etc)
* active haematooncological diseases
* HIV positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy subjects
  2. Patients with invasive candidiasis/Candida sepsis
  3. Patients with sepsis and bacteremia
  4. ICU Patients without infectious disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Biomarkers indicating or excluding invasive Candidiasis | through study completion, an average of 2 years
  Automated (1→3) ß- D- Glucan tests (pg/ml) DNA in serum blood samples (quantity and sequences) pathogen recognition receptors (% of cells as assessed by FACS analysis) serum markers like IL-1, IL-2, IL-6, IL-10, IL-12, IL-17A, IL-17F, IL-22, IL-23, Tryptophan, Kynurenine (quantity) composition of indigenous microbiota of gastrointestinal and lower respiratory tract and skin (comparison of detection rates and abundances of different classes or genera)

SECONDARY OUTCOMES:
Risk factors for Invasive Candidiasis | through study completion, an average of 2 years
  Risk factors as described in previous literature, e.g. Eggimann, Lancet Infect Dis 2003; 3: 685-702

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krause, MD, Principal Investigator — Section of Infectious Diseases and Tropical Medicine, Dpt of Internal Medicine, Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Stmk, Austria

IPD SHARING:
Plan to Share IPD: No